CLINICAL TRIAL: NCT02089698
Title: Mini-flared Kelman Tip and Reverse Tip With Torsional Phaco: Prospective Randomized Comparative Study
Brief Title: Parameters of 2 Phaco Tips Designs in Torsional Phacoemulsification
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Oftalmologico de Brasilia (Other)
Responsible Party: Principal Investigator, PATRICK FRENSEL DE MORAES TZELIKIS, Principal Investigator, Hospital Oftalmologico de Brasilia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014.03
Record Dates: First submitted 2014-03-12; First posted 2014-03-18 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Cataract
Keywords: Kelman tip; Mini-flared; phacoemulsification; cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reversed tip (Active Comparator): Reversed Kelman tip
  Interventions: Device: Mini-flared
- Mini-flared (Experimental): Mini-flared Kelman tip
  Interventions: Device: Reversed tip

INTERVENTIONS:
Device: Mini-flared — Mini-flared Kelman tip
  Arms: Reversed tip
Device: Reversed tip — Reversed Kelman tip
  Arms: Mini-flared

SUMMARY:
To compare the efficiency of surgical procedures using 2 phaco tip designs in torsional phacoemulsification using the bevel-down technique.

DETAILED DESCRIPTION:
In this prospective, comparative, masked study, patients will be randomly assigned to have torsional coaxial microincision cataract surgery using either the mini-flared 45-degree Kelman tip or reversed mini-flared 30-degree Kelman tip. Clinical measurements will include preoperative and 3-month postoperative corrected distance visual acuity (CDVA), endothelial cell counts (ECC) and preoperative and 1-day postoperative central corneal thickness (CCT). Intraoperative measurements will include phaco time, torsional time, aspiration time, case time, cumulative dissipated energy (CDE) and balanced salt solution volume (BSS).

The study was performed according to established ethical standards for clinical research Institutional Review Board (IRB) of the University of Sao Paulo in Brazil, conducted between November 2010 and February of 2011. All surgeries will be performed at the University of Sao Paulo. Physicians conducting postoperative evaluation will not have access to patients' medical records. Exclusion criteria will be previous ocular surgery, central endothelial cell count less than 2000 cells/mm2, glaucoma or intraocular pressure greater than 21 mmHg, amblyopia, retinal abnormalities, steroid or immunosuppressive treatment and connective tissue diseases. Enrolled patients who have complicated cataract surgery (eg, posterior capsule rupture, vitreous loss, or an intraocular lens not placed in the capsular bag) will be subsequently excluded.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 40 years with age-related cataract, and a normal ophthalmologic examination besides senile cataract.

Exclusion Criteria:

* Previous ocular surgery, central endothelial cell count less than 2000 cells/mm2, glaucoma or intraocular pressure greater than 21 mmHg, amblyopia, retinal abnormalities, steroid or immunosuppressive treatment, connective tissue diseases, or an allergy or hypersensitivity to NSAIDs. Enrolled patients who had complicated cataract surgery (eg, posterior capsule rupture, vitreous loss, or an intraocular lens not placed in the capsular bag) were subsequently excluded

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-09; Primary Completion 2013-09 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Early Treatment Diabetic Retinopathy (ETDRS) visual acuities | 90 days

SECONDARY OUTCOMES:
Phaco time used | 1 day, 90 days

OTHER OUTCOMES:
Cumulative dissipated energy (CDE) required | 1 day, 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Patrick F Tzelikis, MD, PhD, Principal Investigator — Hospital Oftalmologico de Brasilia
Locations (1):
- Hospital Oftalmologico de Brasília, Brasília, Federal District, Brazil

REFERENCES:
- [Result] Vargas LG, Holzer MP, Solomon KD, Sandoval HP, Auffarth GU, Apple DJ. Endothelial cell integrity after phacoemulsification with 2 different handpieces. J Cataract Refract Surg. 2004 Feb;30(2):478-82. doi: 10.1016/S0886-3350(03)00620-5. PMID 15030845
- [Result] Payne M, Georgescu D, Waite AN, Olson RJ. Phacoemulsification tip vacuum pressure: Comparison of 4 devices. J Cataract Refract Surg. 2006 Aug;32(8):1374-7. doi: 10.1016/j.jcrs.2006.02.066. PMID 16863978
- [Result] Frohn A, Dick HB, Fritzen CP. Corneal impact of ultrasound and bevel position in phacoemulsification. J Cataract Refract Surg. 2002 Sep;28(9):1667-70. doi: 10.1016/s0886-3350(02)01306-8. PMID 12231329